CLINICAL TRIAL: NCT03797157
Title: Nordic Study on Human Milk Fortification in Extremely Preterm Infants: a Randomized Controlled Trial
Brief Title: Human Milk Fortification in Extremely Preterm Infants
Acronym: N-forte
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thomas Abrahamsson, MD, PhD (Other)
Collaborators: Sahlgrenska University Hospital (Other); Region Uppsala (Unknown); Vasterbottens lans landsting (Unknown); Prolacta Bioscience (Industry); Region Stockholm (Other Government)
Responsible Party: Sponsor-Investigator, Thomas Abrahamsson, MD, PhD, Principal Investigator, MD PhD, Ostergotland County Council, Sweden
Organization: Ostergotland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RegionOstergotland
Record Dates: First submitted 2018-12-17; First posted 2019-01-09 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Necrotizing Enterocolitis; Sepsis; Mortality
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H2MF (Experimental): Human milk-based breast milk fortifier
  Interventions: Dietary Supplement: H2MF
- Standard fortifier (Active Comparator): Standard care: bovine milk-based breast milk fortifier
  Interventions: Dietary Supplement: Bovine milk-based fortifier

INTERVENTIONS:
Dietary Supplement: H2MF — H2MF is a human milk-based breastmilk fortifier for preterm infants
  Arms: H2MF
Dietary Supplement: Bovine milk-based fortifier — Bovine milk-based fortifier is the standard breast milk fortifier in Sweden
  Arms: Standard fortifier

SUMMARY:
This is a randomised controlled multi-centre trial comparing the effect of diet supplementation of a human breast milk-based nutrient fortifier (H2MF®) with standard bovine protein-based nutrient fortifier in 222 extremely preterm infants (born before gestational week 28+0) exclusively fed with human breast milk (own mother´s milk and/or donor milk). The infants will be randomised to receive either the human breast-milk based H2MF® or the standard bovine protein-based nutrient fortifier when oral feeds have reached <100 ml/kg/day.

The randomised intervention, stratified by centre, will continue until the target gestational week 34+0. The infant must not be fed with formula during the intervention period. The allocation will be concealed before inclusion, but after randomisation the study is not blinded.

Primary endpoint of the intervention is the composite variable necrotizing enterocolitis (NEC), sepsis and mortality.

The enrolled infants are characterised with clinical data including growth, feeding intolerance, use of enteral and parenteral nutrition, treatment, antibiotics and complications collected daily in a study specific case report form from birth until discharge from the hospital (not longer than gestational week 44+0). A follow up focusing on neurological development, growth and feeding problems will be performed at 2 years of age (corrected) and 5.5 years of age.

DETAILED DESCRIPTION:
This is a randomised controlled multi-centre trial comparing the effect of diet supplementation of a human breast milk-based nutrient fortifier (H2MF®) with standard bovine protein-based nutrient fortifier in 222 extremely preterm infants (born before gestational week 28+0) exclusively fed with human breast milk (own mother´s milk and/or donor milk). The infants will be randomised to receive either the human breast-milk based H2MF® or the standard bovine protein-based nutrient fortifier when oral feeds have reached <100 ml/kg/day. If fortification with extra enteral lipids is needed during the intervention period, the infants receiving H2MF® will be supplemented with the human milk-based Prolact CR®, while the infants receiving standard bovine protein-based fortification will be supplemented with the standard lipid products used at the unit. The study subject will be enrolled at level III neonatal intensive care unit (NICU)s. Only infants with a home clinic with the logistics to maintain the intervention until gestational week 34+0 will be included.

The randomised intervention, stratified by centre, will continue until the target gestational week 34+0. The infant must not be fed with formula during the intervention period. The allocation will be concealed before inclusion, but after randomisation the study is not blinded. It would not be possible to prescribe the fortifier and prepare of the breast milk in a blinded fashion, since the fortifiers are not exactly equal in nutrient content and also look different. Instead the assessment of several of the outcomes will be made blinded, such as the assessment of X-ray images in NEC cases.

The enrolled infants are characterised with clinical data including growth, feeding intolerance, use of enteral and parenteral nutrition, treatment, antibiotics and complications collected daily in a study specific case report form from birth until discharge from the hospital (not longer than gestational week 44+0). A follow up focusing on neurological development, growth and feeding problems will be performed at 2 years of age (corrected) and 5.5 years.

Since it is often difficult to distinguish between the diagnoses of NEC and sepsis, and their clinical consequences, the investigator's primary endpoint of the intervention is the composite variable NEC, sepsis and mortality. Secondary endpoints are feeding intolerance and other severe complication such as Bronchopulmonary dysplasia (BPD), Retinopathy of prematurity (ROP) and neurological impairment. Stool, urine and blood samples are also collected for microbiology, metabolomic and immunology analysis in order to study underlying mechanisms. Health economic analyses will be made to evaluate the costs and benefits of an introduction of human milk-based fortifier in NICUs in the Nordic countries.

Analyses will be conducted using an intention to treat approach. An evaluation will be performed when 20 infants have been included to evaluate feasibility and make it possible to adjust the protocol for the remaining part of the study. Safety analyses will be performed by an independent data and safety monitoring board (DSMB) when 50, 100 and 150 infants have been included. A sample size re-estimation will be made by an independent statistician when 150 infants have been included. Thus, the definitive sample size might be increased (never decreased) based on this interim analysis. The study can be terminated before 322 infants have been enrolled based on a decision of the sponsor and the DSMB, if the primary outcome is significantly lower (with a significance level <0.001) in the H2MF® than in the standard fortification group in the interim analysis made after 150 infants have completed the neonatal period. The study subject will be enrolled at level III NICUs in the Nordic Countries. All study subjects will be followed during the neonatal period until discharge (not longer than gestational week 44+0) and also be included in a follow up at 2 and 5.5 years of age based on the national follow up program for extremely preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth 22+0-27+6: based on prenatal ultrasonography.
* Enteral feeds < 100 mL/kg/day at the day of randomisation.
* Written informed consent from the legal guardians of the infant.
* The home clinic of the infant has the logistics of maintaining the intervention until gestational week 34+0

Exclusion Criteria:

* Lethal or complicated malformation known at the time of inclusion
* Chromosomal anomalies known at the time of inclusion
* No realistic hope for survival at the time of inclusion
* Gastrointestinal malformation known at the time of inclusion
* Abdominal surgery before the time of inclusion
* Participation in another intervention trial aiming at having an effect on growth, nutrition, feeding intolerance or severe complications such as NEC and sepsis
* Infants having nutrient fortifier or formula prior to randomisation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of the composite of necrotizing enterocolitis, culture-proven sepsis and mortality | From birth until discharge from hospital (but not longer than gestational week 44+0)
  An infant should have had any of these diagnoses to fulfil the criterion

SECONDARY OUTCOMES:
The incidence of the composite of necrotizing enterocolitis and culture-proven sepsis | From birth until discharge from hospital (but not longer than gestational week 44+0)
  An infant should have had any of these diagnoses to fulfil the criterion
The incidence of the composite of necrotizing enterocolitis culture-proven sepsis, bronchopulmonary dysplasia, retinopathy of prematurity and mortality (Mortality and morbidity index) | From birth until discharge from hospital (but not longer than gestational week 44+0)
  An infant should have had any of these diagnoses to fulfil the criterion
Time to reach full enteral feeds | From birth until discharge from hospital (but not longer than gestational week 44+0)
  The day of life the infant has received at least 150 mL/kg enteral feeds
Number of feeding interruptions | From birth until discharge from hospital (but not longer than gestational week 44+0)
  Number of days feedings held for ≥12 hours or feeds reduced by >50% (ml/kg/d) not due to a clinical procedure or transitioning to the breast
Numbers of days with parenteral nutrition | From birth until discharge from hospital (but not longer than gestational week 44+0)
  Number of days of parental amino acid and/or lipid infusion. Only days when the enteral feed <150mL/kg/day should be included
Number of large gastric aspirates per day | From birth until discharge from hospital (but not longer than gestational week 44+0)
  ≥100% pre-feed volume (2 hours feeding volume if continuous feeding). Lower limit=2 ml/kg.
Stool frequency | From birth until discharge from hospital (but not longer than gestational week 44+0)
Time to regain birth weight | From birth until discharge from hospital (but not longer than gestational week 44+0)
Change in head circumference in centimeters | At 7, 14, 21 and 28 days, the end of intervention (gestational week 34+0), gestational week 36+0, at discharge from neonatal ward (or at gestational week 44+0, whatever comes first) and at 2 years of age (corrected) and 5.5 years of age (uncorrected).
Change in weight in gram | At 7, 14, 21 and 28 days, the end of intervention (gestational week 34+0), gestational week 36+0, at discharge from neonatal ward (or at gestational week 44+0, whatever comes first) and at 2 years of age (corrected) and 5.5 years of age (uncorrected).
Change in length in centimeters | At 7, 14, 21 and 28 days, the end of intervention (gestational week 34+0), gestational week 36+0, at discharge from neonatal ward (or at gestational week 44+0, whatever comes first) and at 2 years of age (corrected) and 5.5 years of age (uncorrected).
The mortality incidence | From birth until discharge from hospital (but not loner than gestational week 44+0)
The incidence of necrotising enterocolitis: Bell´s stage II-III | From birth until discharge from hospital (but not loner than gestational week 44+0)
The incidence spontaneous intestinal perforation | From birth until discharge from hospital (but not loner than gestational week 44+0)
The incidence of abdominal surgery | From birth until discharge from hospital (but not loner than gestational week 44+0)
The incidence culture-proven sepsis | From birth until discharge from hospital (but not loner than gestational week 44+0)
The incidence of suspected sepsis, not culture-proven | From birth until discharge from hospital (but not loner than gestational week 44+0)
The incidence of pneumonia | From birth until discharge from hospital (but not loner than gestational week 44+0)
  Pathological X-ray confirmed by an independent radiologist, need of increased respiratory support/oxygen and laboratory inflammatory response
The incidence of bronchopulmonary dysplasia | At gestational week 36+0
  Need of extra oxygen, continuous positive air pressure (CPAP) or ventilator at gestational week 36+0
The incidence of retinopathy of the prematurity | From birth until gestational week 42+0
  Classified into stage I-V. The diagnosis is set after gestational week 42+0
The incidence of intraventricular haemorrhage | From birth until discharge from hospital (but not loner than gestational week 44+0)
  Classified into grade I-IV according to Papile
The incidence of periventricular leukomalacia | From birth until discharge from hospital (but not loner than gestational week 44+0)
  Criteria according to de Vries
Number of days with intensive care | From birth until discharge from hospital (but not loner than gestational week 44+0)
  Need of respirator or CPAP until discharge (not later than gestational week 44+0).
Length of stay at the hospital | From birth until discharge from hospital (but not loner than gestational week 44+0)
  Gestational week and day at discharge (not later than gestational week 44+0).
Length of need of feeding tube | From birth until discharge from hospital (but not loner than gestational week 44+0)
  Gestational week and day when the infant does not need it anymore (not later than gestational week 44+0)
Neurocognitive development at 2 years | At 2 years of age
  Bayleys III, PARCA-R (Parental Report of Children´s Abilities-Revised) and ASQ-3 (Ages and stages questionnaire)
Prevalence of cerebral palsy at 2 years | At 2 years of age
Prevalence of epilepsy at 2 years | At 2 years of age
Prevalence of squint and/or impaired vision at 2 years | At 2 years of age
Prevalence of impaired hearing at 2 years | At 2 years of age
The number of infants needing extra oxygen and/or ventilatory support after discharge from the hospital at the neonatal period | From gestational week 44 until 2 years of age
The incidence of wheeze and/or asthma | From birth until 2 years of life
The incidence of severe infections after discharge from the neonatal unit | From gestational week 44 until 2 years of age
The number of infants needing feeding tube after discharge from the hospital at the neonatal period | From gestational week 44 until 2 years of age
The number of infants needing extra nutritional support after discharge from the hospital at the neonatal period | From gestational week 44 until 2 years of age
The prevalence of neurocognitive development at 5.5 years | At 5.5 years of age
  Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI-IV TM) and Movement ABC-2: the total scale points as well as the points of sub scales (motor, cognitive, language) will be presented. The prevalence of infants with a realist below 2 standard deviations will be defined to have mental retardation.
The prevalence of cerebral palsy at 5.5 years | At 5.5 years of age
The prevalence of epilepsy at 5.5 years of age | At 5.5 years of age
The prevalence of squint and/or impaired vision at 5.5 years of age | At 5.5 years of age
The prevalence of children with impaired hearing at 5.5 years of age | At 5.5 years of age
The prevalence of wheeze and/or asthma at 5.5 years of age | At 5.5 years of age
Microbiome composition in stool samples | At 1, 2, 3 and 4 weeks of age and gestational week 36+0
  The relative abundance and diversity of microbial taxa will be analyses with next generation sequencing and be related till the study intervention
Levels of subclasses of T and B cells and granulocytes in blood samples | At 1, 2 and 4 weeks of age and gestational week 36+0
  T helper subsets (TH1, Th2, TH17, Treg), T cells subsets associated with the intestinal mucosa (gamma/delta-T cells, MAIT cells) and neutrophils will be assessed using masscytometry
Levels of immune markers in plasma | At 1, 2 and 4 weeks of age and gestational week 36+0
  Pre planned analyses are anti-inflammatory (e.g. IL-10) and proinflammatory (e.g. TNF) cytokines and chemokines (e.g. CXCL11, CCL18).
Levels of growth factors in plasma samples | At 1, 2 and 4 weeks of age and gestational week 36+0
  The levels of growth factors such as IGF-1 and the associated IGFBP-3 will be analysed.
Levels of lipids in plasma samples | At 1, 2 and 4 weeks of age and gestational week 36+0
  Fatty acids in plasma
Levels of neurotransmitters in plasma samples | At 1, 2 and 4 weeks of age and gestational week 36+0
  Neurotransmitters such as GABA and serotonin in plasma
Levels of metabolic peptides in urine samples | At 1, 2, 3 and 4 weeks of age and gestational week 36+0
  Metabolic peptide will be measured with proton nuclear magnetic resonance spectroscopy (NMR), liquid chromatography (LC) and mass spectroscopy couple to gas chromatography (GC-MC).
Levels of markers of central nervous system (CNS) damage in plasma samples | At 1, 2 and 4 weeks of age and gestational week 36+0
  Markers of CNS damage such as neurofilament light protein will be measured in plasma
Levels of proteins in breast milk samples | At 1, 2, 3 and 4 weeks of age and gestational week 36+0
  Protein composition will be measured with multiplex methods
Levels of human milk oligosaccharides in breast milk samples | At 1, 2, 3 and 4 weeks of age and gestational week 36+0
  The levels of human milk oligosaccharides will be measured with high-performance anion-exchange chromatography with pulsed amperometric detection.
Health care costs | From birth until discharge from hospital (but not loner than gestational week 44+0)
  The number of days at each level of care will be recorded until discharge from the hospital (not longer than gestational week 44+0). The cost will be calculated by multiplying the number of days at each level of care by the average cost

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Abrahamsson, MD, PhD, Principal Investigator — Region Östergötland
Locations (5):
- Sweden (5):
  - Queen Silvia Children´s Hospital, Gothenburg
  - Crown Princess Victoria Children´s Hospital, Linköping
  - Karolinska Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Barnsjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen GB, Domellof M, Ahlsson F, Elfvin A, Naver L, Abrahamsson T. Effect of human milk-based fortification in extremely preterm infants fed exclusively with breast milk: a randomised controlled trial. EClinicalMedicine. 2024 Jan 2;68:102375. doi: 10.1016/j.eclinm.2023.102375. eCollection 2024 Feb. PMID 38545091
- [Derived] Jensen GB, Ahlsson F, Domellof M, Elfvin A, Naver L, Abrahamsson T. Nordic study on human milk fortification in extremely preterm infants: a randomised controlled trial-the N-forte trial. BMJ Open. 2021 Nov 23;11(11):e053400. doi: 10.1136/bmjopen-2021-053400. PMID 34815288

DOCUMENTS (3):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03797157/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03797157/SAP_001.pdf
  • Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03797157/ICF_002.pdf